CLINICAL TRIAL: NCT06990113
Title: Effect of Three-dimensional Lumbar Myofascial Release With Motor Control Training on Back Perception and Pain in Patients With Lumbar Radiculopathy
Brief Title: Three-dimensional Lumbar Myofascial Release and Motor Control in Lumbar Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005789
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: The patients were randomly divided into two equal groups; Study group (16 patients): received three dimensional lumbar myofascial release with motor control training, and conventional treatment. Control group (16 patients): received conventional treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): received three dimensional lumbar myofascial release with motor control training, and conventional treatment
  Interventions: Other: three dimensional lumbar myofascial release; Other: conventional treatment.
- control group (Experimental): received conventional physical therapy modalities, including electrotherapy and flexibility treatment
  Interventions: Other: conventional treatment.

INTERVENTIONS:
Other: three dimensional lumbar myofascial release — Three-dimensional (3D) MFR is a novel approach toward reducing fascial restrictions. It recognizes that fascia exists not only in a linear plane but also in complex multidirectional networks throughout the body.
  Other Names: (3D) MFR
  Arms: study group
Other: conventional treatment. — conventional treatment, including selected physical therapy, flexibility exercise for the back, static back and abdomen exercises, and electrotherapy

SUMMARY:
to investigate The Efficacy of three-dimensional lumbar myofascial release with motor control training on back perception and pain in lumbar radiculopathy Patients with lumbar radiculopathy demonstrate impairments in function and range of motion to deficits in patient's quality of life.

DETAILED DESCRIPTION:
PURPOSE: to investigate The Efficacy of three-dimensional lumbar myofascial release with motor control training on back perception and pain in lumbar radiculopathy Patients with lumbar radiculopathy demonstrate impairments in function and range of motion to deficits in patient's quality of life.

HYPOTHESES: It will be hypothesized that there will be no statically Effect of three dimensional lumbar myofascial release with motor control training on back perception and pain in lumbar radiculopathy RESEARCH QUESTION: Is there an Effect of three-dimensional lumbar myofascial release with motor control training on back perception and pain in lumbar radiculopathy

ELIGIBILITY:
Inclusion Criteria:

* Their ages range from 35 to 50 years.
* Both sex
* Unilateral lumbar radiculopathy for more than 6 months.
* Normal body mass index (18.5 - 24.99Kg/m2).

Exclusion Criteria:

* • Any other musculoskeletal disorders of the spine or upper extremity

  * Patients with any other Neurological deficits, psychiatric disease lumbar myelopathy, Cognitive problems, vertebral fractures and previous history of spine or lumbar surgery.
  * Clinical instability, recent trauma
  * Structural abnormalities of the spine, osteoporosis, and spasmodic torticollis.
  * Inflammatory or other specific disorders of spina such as ankylosing spondylitis and rheumatoid arthritis

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Fremantle Back Awareness Questionnaire | four weeks
  The Fremantle Back Awareness Questionnaire (FreBAQ) has been found to possess adequate psychometric properties in low back pain (LBP) patients worldwide
Oswestry Low Back Pain Disability Questionnaire | four weeks
  The Oswestry Disability Index (ODI) a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain

SECONDARY OUTCOMES:
pressure pain algometer | four weeks
  Algometers are designed to quantify and document levels of tenderness via pressure pain threshold measurement and pain sensitivity via pressure pain tolerance measurement.
visual analog scale | four weeks
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Lama Saad El-Din Mahmoud, Al Jīzah, Select State, Egypt